CLINICAL TRIAL: NCT02976649
Title: Proposal of a Score to Detect the Need for Postoperative Intensive Care Unit Admission After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Walid Nofal, Lecturer of Anesthesiology, Ain Shams University
Other Study IDs: FMASU R 19/2016
Record Dates: First submitted 2016-11-22; First posted 2016-11-29 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Bariatric Surgery Procedures
Keywords: Morbid obesity; Bariatric surgery; Multi-dimensional score
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to propose a multi-dimensional score to predict those patients undergoing bariatric surgeries who will be in need for postoperative ICU admission.

DETAILED DESCRIPTION:
A multi-dimensional score of 7 risk factors was proposed which may help in identifying morbidly obese patients undergoing bariatric surgeries who will need admission to a critical care unit postoperatively for follow up.

ELIGIBILITY:
Inclusion Criteria:

* patients who have been operated upon for either laparoscopic gastric sleeve or laparoscopic gastric bypass during the period from January to June 2016.

Exclusion Criteria:

* Patients were excluded in case of postoperative surgical complications, conversion to open surgery or in case of redo.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbid obese patients who have been operated upon for either laparoscopic gastric sleeve or laparoscopic gastric bypass.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Creation of a multi-dimensional score for the need of post-bariatric surgery ICU admission | Through study completion, an average of six months.

CONTACTS AND LOCATIONS:
Overall Officials: Walid H. Nofal, MD, Principal Investigator — Anesthesiology department, Faculty of Medicine, Ain Shams University
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided